CLINICAL TRIAL: NCT06833515
Title: A Paradigm Change in Root Canal Preparation: Can Reciprocal Files Be Used Alone?
Brief Title: The Effect of Using Reciprocal Files Alone and with Different Files on Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Nezif Celik, assistant professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRÜ-DHF-END-NC-02
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain; Chronic Apical Periodontitis of Pulpal Origin
Keywords: rotary; reciproc; mode; pain; periodontitis
MeSH Terms: conditions — Pain, Postoperative; Pain; Periodontitis

STUDY DESIGN:
Intervention Model Description: experimental groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- one flare+wave one gold glider+wave one gold (Active Comparator): Using a #10K-type stainless-steel file, the operator will establish the working length 0.5 mm short of the apex indicated by the Root ZX Mini apex locator and will confirm it on periapical radiograph. The operator then will irrigate the root canals with 2 mL of 5%NaOCl . Teeth in this group will first be shaped in rotational mode using One Flare. Then, they will be shaped using WaveOne Gold Glider and WaveOne in reciprocal mode. After the treatment, the patient's pain score will be recorded.
  Interventions: Other: one flare+wave one gold glider+wave one gold
- waveone gold glider+waveone gold (Active Comparator): Using a #10K-type stainless-steel file, the operator will establish the working length 0.5 mm short of the apex indicated by the Root ZX Mini apex locator and will confirm it on periapical radiograph. The operator then will irrigate the root canals with 2 mL of 5%NaOCl. this group teeth will be operated using reciprocal motion with waveone gold glider and waveone gold. After the treatment, the patient's pain score will be recorded.
  Interventions: Other: wave one gold glider+wave one gold
- waveone gold (Active Comparator): Using a #10K-type stainless-steel file, the operator will establish the working length 0.5 mm short of the apex indicated by the Root ZX Mini apex locator and will confirm it on periapical radiograph. The operator then will irrigate the root canals with 2 mL of 5%NaOCl. this group teeth will be operated using reciprocal motion with wave one gold. After the treatment, the patient's pain score will be recorded.
  Interventions: Other: wave one gold
- 15K-type stainless-steel hand file (Placebo Comparator): The operator will prepare the glide path using a
  * 15K-type stainless-steel hand file with push-pull motion. On sensing resistance, the file was withdrawn, recapitulation will performe with a #10K-type stainless-steel file, and debris will removed by irrigating the canals with 5% NaOCl. The operator repeated this procedure until the
  * 15K-file reached the complete working length.
  Interventions: Other: 15K-type stainless-steel hand file

INTERVENTIONS:
Other: one flare+wave one gold glider+wave one gold — In this clinical study, the teeth will first undergo coronal shaping with the One Flare file. Then, the glide path and final shaping will be performed in reciprocal mode with reciprocal files.
  Arms: one flare+wave one gold glider+wave one gold
Other: wave one gold glider+wave one gold — In this group, only the glide path and final shaping will be performed using reciprocal files, without coronal shaping.
  Arms: waveone gold glider+waveone gold
Other: wave one gold — In this group, shaping will be performed using only a reciprocating file, without coronal shaping and glide path preparation.
  Arms: waveone gold
Other: 15K-type stainless-steel hand file — The operator prepared the glide path using a #15K-type stainless-steel hand file with push-pull motion. On sensing resistance, the file was withdrawn, recapitulation was performed with a #10K-type stainless-steel file, and debris was removed by irrigating the canals with 5% NaOCl. The operator repeated this procedure until the #15K-file reached the complete working length
  Arms: 15K-type stainless-steel hand file

SUMMARY:
This study aims to investigate the effects of using the Wave One Gold file alone and in combination with different files on postoperative pain in patients with asymptomatic apical periodontitis. The results of the study may provide important insights into the impact of these file systems on postoperative pain. . The main questions it aims to answer are:

It will also reveal whether reciprocating files can be used alone or not.

Participants will:

Go under treatment with different shaping protocols The researchers will shape using only the Wave One gold file in the first group.

In the second group, they will first perform coronal shaping with the One Flare file and then complete the final shaping with the Wave One Gold file In the third group, coronal shaping will first be performed with the One Flare, followed by working length shaping with the Wave One Gold glider file, and the final shaping will again be completed with the Wave One file. For sham group Using a #10K-type stainless-steel file, the operator will establish the working length 0.5 mm short of the apex indicated by the apex locator and will confirm it on periapical radiograph. The operator will prepare the glide path using a #15K-type stainless-steel hand file with push-pull motion.On sensing resistance, the file will withdraw.

recapitulation was performed with a #10K-type operator then will irrigate the root canals with 2 mL of 5%NaOCl . Then, they will be shaped using WaveOne Gold Glider and WaveOne in reciprocal mode. After the treatment, the patient's pain score will be recorded.

They will Visit the clinic three days later Keep avisual analogue scala of their symptoms and than compare different shaping protocols

DETAILED DESCRIPTION:
Randomization The names of systems will write on the papers, the papers will fold, and these papers will placed into a dark box, which cannot be seen from theoutside. Before each treatment, the clinical assistant chose a paper randomly from the dark box and the system written in that paper will applied to the patient.

Treatment Protocol A single operator will performe root canal treatment for all the patients in 2 sessions. The operator will administer local anesthesia with 2 mL of 4 articaine and 1:100,000 epinephrine (Ultracain DS Fort; Aventis _ Ilaç A.S x, Istanbul, Turkey) 10 minute before the procedure. Then, the tooth of interest will isolate using a rubber dam. Caries or coronal restorations will remove completely, and the endodontic access cavity will open using diamond fissure burs(Diatech,Diamant AG, Switzerland) under water-cooled conditions. After negotiating the root canal orifices, the apical patency of the teeth wil checked

The study will be examined wave one gold with/without one flare and wave one gold glider. First, in the first group, the Wave One Gold file will be used as a single-file system according to the manufacturer's usage instructions. In the second group, the One Flare file will be used first, and the final shaping will be done with the Wave One Gold file. In the third group, the One Flare file will be used first, followed by the Wave One Gold glider, and the final shaping will be performed with the Wave One Gold file.

As a rinsing protocol, each file change will be followed by a rinse with 2 mL of using a side-perforated 30 G needle . In the final rinse, 10 mL of 17% EDTA and 10 mL of 2.5% NaOCl will be activated ultrasonically.

Later, patients will be informed about the visual analog scale (VAS). Patients will be called for a check-up three days later. The evaluation scores of the patients and their use of painkillers will be noted.

Statistical analysis A sample size calculation was performed using the G∗Power software (G∗Power 3.1.9.7; Heinrich-Heine Universität, Düsseldorf, Germany) based on a 0.05 type I error, 80% power, and an effect size of 0.25. According to Cohen, the minimum sample size required to detect differences in postoperative pain intensity among 4 study groups at 3 time points would be 36. Since this study was analyzed using non-parametric methods, a decision was made to include 42 patients (36 * 1.15 = 42) as suggested by Lehmann, with 42 patients allocated to each group; this number was sufficient to ensure statistical significance. In comparing multiple group contrasts and repeated measurements, ANOVA test will be used. The Shapiro-Wilk test will be employed to check for normal distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* Adult, systemically healthy patients aged18-65years(category:AmericanSocietyof Anesthesiologists class 1.
* Patients diagnosed with symptomatic reversible pulpitis and having mandibular first and second premolar teeth without percussion pain.
* Teeth with prolonged response to the coldpulp test (Endo-Frost, Coltene-Whaledent, Allstetten, Switzerland) (teeth where pain persists for a long time after stimulus removal)
* Teeth with normal periapical appearance(periapical index 2), a single root canal andaroot canal inclination less than 20° on a parallel periapical radiograph
* Teeth with moderately sharp spontaneous pain (preoperative visual analog scale [VAS] score 4-6)
* Teeth where number 10 K files can reach and fit the working lenght
* Patients who were able to understand the informed consent form and pain recording scales used in the study were included

Exclusion Criteria:

* Patients who are pregnant and lactating
* Patients who received analgesics or anti inflammatory drugs in the last 12 hours and antibiotics for the last 1 month
* Patients with severe periodontal defect or deep periodontal pocket (probing depth.3 mm)and poor oral hygiene
* Teeth too broken down, difficult to isolate with rubber dam
* Teeth without occlusal contact
* Presence of multiple teeth requiring treatment, a previous treatment history and an open apex
* Teeth with calcified root canal, root resorption, crown and/or root fracture, multiple root canals, post, and sinus tract were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
visual analoge scala | 24-48-72 hours
  it contains 5 different images correlated with severity of pain with 10 numeric levels of pain. Minimum value of pain is 1 while the highest value is 10. 10 is a worse value of pain than 1.

CONTACTS AND LOCATIONS:
Overall Officials: tolga han edebal, PhD, Study Chair — HARRAN UNİVERSTY
Locations (1):
- Nezif Çelik, Karaköprü, Şanlıurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No